CLINICAL TRIAL: NCT02958124
Title: Early Mobilization: Evaluation of Feasibility and Security in Pediatric Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: MobpediaSIP
Record Dates: First submitted 2016-09-14; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Cardio-Respiratory Distress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the feasibility and the security of early mobilization of infants in pediatric intensive care.

ELIGIBILITY:
Inclusion Criteria:

* cardiorespiratory stability
* between 24 and 48h post admission

Exclusion Criteria:

* Thorax open
* ECLS
* High frequency oscillatory ventilation

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients admitted in pediatric intensive care unit that respond to eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory parameters assessed by monitoring | up to 1 hour
  cardiac frequency, respiratory frequency, blood pressure

SECONDARY OUTCOMES:
EDIN scale (tool for assessing prolonged pain in preterm and newborns) | 5 minutes before mobilization
EDIN scale (tool for assessing prolonged pain in preterm and newborns) | up to 1 hour
COMFORT-BEHAVIOR scale (to measure the amount of stress of ventilated infants in a pediatric intensive care unit) | 5 minutes before mobilization
COMFORT-BEHAVIOR scale (to measure the amount of stress of ventilated infants in a pediatric intensive care unit) | up to 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

REFERENCES:
- [Derived] Piva TC, Ferrari RS, Schaan CW. Early mobilization protocols for critically ill pediatric patients: systematic review. Rev Bras Ter Intensiva. 2019 Jun 10;31(2):248-257. doi: 10.5935/0103-507X.20190038. PMID 31215603